CLINICAL TRIAL: NCT00995007
Title: A Randomized Phase II Trial of Vandetanib (ZD6474) in Combination With Carboplatin Versus Carboplatin Alone Followed by Vandetanib Alone in Adults With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine E. Warren, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090222; 09-C-0222
Record Dates: First submitted 2009-10-10; First posted 2009-10-14 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Mixed Oligoastrocytoma
Keywords: Brain Tumor; Chemotherapy; Antiangiogenesis; Radiation; Progression; Glioma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms; Disease Progression; Glioma | interventions — vandetanib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Active Comparator): Sequential Group (carboplatin followed by vandetanib)
  Interventions: Drug: ZD6474 (Vandetanib); Drug: Carboplatin
- Group 1 (Active Comparator): Combo Group (both drugs together)
  Interventions: Drug: ZD6474 (Vandetanib); Drug: Carboplatin

INTERVENTIONS:
Drug: ZD6474 (Vandetanib) — Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
Drug: Carboplatin — Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.

SUMMARY:
Background:

* Growth of new blood vessels (angiogenesis) provides many tumors, including brain tumors, with needed nutrients and oxygen for cancer cells to survive. One possible treatment for different kinds of cancer involves treatment with drugs that slow or stop angiogenesis and prevent further tumor growth.
* Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
* Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.

Objective:

- To determine the safety and effectiveness of vandetanib and carboplatin, given together or sequentially, against recurrent high-grade gliomas.

Eligibility:

- Adults diagnosed with a malignant glioma who have received standard treatments that no longer appear to be effective.

Design:

* Patients will be assigned to one of two groups. Group 1 patients (combination group) will receive oral vandetanib for 28 days and intravenous (IV) carboplatin (once at the beginning of the 28-day cycle). Group 2 patients (sequential group) will receive IV carboplatin alone (once at the beginning of the 28-day cycle) and then oral vandetanib (300 mg daily) for 28 days if the tumor grows or the patient develops unacceptable carboplatin toxicity.
* Treatment will continue in 28-day cycles for 1 year for both groups.
* Patients will undergo a number of tests and procedures during the treatment cycle, including physical examinations, routine laboratory tests, electrocardiograms, and magnetic resonance imaging (MRI) scans
* At the end of 1 year of treatment, patients will be reevaluated for possible continuation of drug therapy.

DETAILED DESCRIPTION:
Background:

In vivo experiments have documented the ability of vandetanib (ZD6474) to inhibit tumor growth in various preclinical tumor models. Given the pronounced neovasculature associated with malignant gliomas, and abundant published data demonstrating the dependence of glioma growth on the maintenance and proliferation of this neovasculature, vandetanib represents a potentially promising new therapeutic approach to these otherwise refractory tumors. Phase II data of vandetanib for recurrent glioblastomas conducted at the National Institutes of Health showed promising activity but responses were usually short-lasting.

Carboplatin has shown activity as monotherapy in the treatment of recurrent malignant gliomas in adults and preclinical data generated at Dr. Fines' laboratory demonstrate additive anti-glioma activity with vandetanib. The safety profile of carboplatin and the preclinical and clinical data supports its use in combination with vandetanib in patients with malignant gliomas.

Vandetanib is also an epidermal growth factor receptor (EGFR) inhibitor and it has been demonstrated that the presence of the EGFRvIII mutant and/or the presence of an intact phosphatase and tensin homolog deleted on chromosome 10 (PTEN) and non-phosphorylated protein kinase B (AKT) predict for a higher likelihood of response to the EGFR inhibitors Tarceva and Iressa.

Objectives:

To establish data regarding the anti-tumor activity of vandetanib in combination with carboplatin and single agent carboplatin and to collect information regarding the spectrum of toxicities.

To determine if the presence of the EGFRvIII mutant and/or the presence of an intact PTEN and non-phosphorylated AKT predict for a higher likelihood of response to vandetanib.

Eligibility:

Patients with histologically proven malignant glioma are eligible for this study.

Design:

Patients will be randomized (1:1) to one of two groups. Patients in group one will be treated with vandetanib (300 mg daily for patients not on enzyme inducing anti-epileptic drugs (EIAEDs) and 400 mg daily for patients on EIAEDs) and with carboplatin (area under the concentration-time curve at steady-state [area under curve (AUC)], 6mg/mL x min) once every 4-week cycle (combination group). Patients in group two will receive carboplatin alone (AUC 6mg/mL x min) once every 4-week cycle. Patients who develop tumor progression or unacceptable toxicity on carboplatin alone (group 2) can then receive single agent vandetanib (300 mg daily for patients not on enzyme inducing anti-epileptic drugs (EIAEDs) and 400 mg daily for patients on EIAEDs) in 4-week cycles (sequential group). A total of 128 evaluable patients will be analyzed. The total accrual ceiling will allow for 74 patients to be enrolled in the glioblastoma multiforme (GBM) stratum and 74 patients in the anaplastic gliomas (AG) stratum (total 148) to factor in replacing those patients who come off treatment prior to cycle 1.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with histologically proven malignant primary gliomas who have progressive disease after radiotherapy will be eligible for this protocol. These include glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), and malignant glioma/astrocytoma NOS.

Patients must have an magnetic resonance imaging (MRI)/computed tomography (CT) scan performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MRI/CT is required. The same type of scan, that is, MRI or CT must be used throughout the period of protocol treatment for tumor measurement.

Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

Patients will be eligible four weeks after surgery if they have recovered from the effects of surgery.

Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/MRI should be done:

* no later than 96 hours in the immediate post-operative period or
* at least 4 weeks post-operatively, and
* within 14 days of registration, and
* on a steroid dosage that has been stable for at least 5 days.

If the 96 hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.

Patients must have failed prior radiation therapy.

All patients or their previously designated durable power of attorney (DPA) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.

Patients must be greater than or equal to 18 years old, and must have a life expectancy greater than 8 weeks.

Patients must have a Karnofsky performance status of greater than or equal to 60.

Patients must be at least six weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide, 3 weeks from procarbazine, and 2 weeks from last vincristine administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents.

Patients must have adequate bone marrow function (white blood cell (WBC) greater than or equal to 3,000/microL, absolute neutrophil count (ANC) greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase 2.5 less than or equal to upper limit of normal (ULN) and bilirubin less than or equal to 1.5 times ULN), and adequate renal function (creatinine less than or equal to 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. Patients must also have serum potassium greater than or equal to 3.5 mg/dL, magnesium greater than or equal to 0.75 mmol/L and calcium levels within normal levels; supplementation is allowed. In cases where the serum calcium is below the normal range, 2 options would be available: 1) the calcium adjusted for albumin is to be obtained and substituted for the measured serum value. Exclusion is to then be based on the adjusted for albumin values falling below the normal limit. 2) Determine the ionized calcium levels. Exclusion is then to be based if these ionized calcium levels are out of normal range despite supplementation. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.

This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

Patients must not be pregnant or nursing, and all patients (both men and women) must be willing to practice birth control during and for 2 months after treatment with vandetanib and/or carboplatin. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition, WCBP patients must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

A 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial entry with corrected QT interval (QTc) less than 480 msec. If a patient has a QT interval corrected for heart rate using Bazett's) QTcB interval > 480 ms on screening ECG, the screening ECG may be repeated twice [at least 24 hours apart] for a total of 3 ECGs. The average QTcB from the 3 screening ECGs must be less than or equal to 480 ms in order for the patient to be eligible for the study).

EXCLUSION CRITERIA:

Patients who, in the view of the treating physician, have significant active hepatic, renal, or psychiatric diseases are ineligible.

Prior treatment with vandetanib.

Prior treatment with platinum-based therapy.

Patients known to have an allergic response to mannitol.

Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease greater than or equal to 2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.

History of arrhythmia (multifocal premature ventricular contractions PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (Common Terminology Criteria for Adverse Events (CTCAE) grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.

QTc prolongation with other medications that required discontinuation of that medication.

Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.

Presence of left bundle branch block (LBBB.)

QTc with Bazett's correction that is unmeasurable, or greater than or equal to 480 msec on screening ECG. (Note: If a subject has a QTc interval greater than or equal to 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than 480 msec in order for the subject to be eligible for the study. Patients who are receiving a drug that has a risk of QTc prolongation excluded if QTc is greater than or equal to 460 msec.

Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes. Drugs listed in Appendix E, Table 2, that in the investigators opinion cannot be discontinued are allowed; however, must be monitored closely with additional ECGs and laboratory assessments of electrolytes to ensure the patients safety.

Concomitant medications that are potent inducers (rifampicin, rifabutin, St. Johns Wort and Enzyme-Inducing Anti-Epileptic Drugs (EIAEDs) of cytochrome P450 3A4 (CYP3A4) function. EIAEDs are allowed.

Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)

Currently active diarrhea that may affect the ability of the patient to absorb the vandetanib or tolerate diarrhea.

Women who are currently pregnant or breast feeding.

Patients known to have a malignancy (other than their malignant glioma) that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except for non-melanoma skin cancer, carcinoma in situ in the cervix or ductal carcinoma in situ).

Invasive procedures defined as follows:

* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to Day 1 (D1) therapy

Patients should not be on anti-platelet medications (aspirin, clopidogrel, ticlopidine, prasugel). Non-steroidal anti-inflammatory drugs should be used with caution if medically necessary.

Restrictions

* Patients who are blood donors should not donate blood during the trial and for 3 months following their last dose of trial treatment.
* Due to the experimental nature of vandetanib, all patients of childbearing potential must be one year post-menopausal, surgically sterile, or using an acceptable method of contraception (oral contraceptives, barrier methods in conjunction with spermicide,

approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) during and continued after the last dose of study medication. Contraceptive use will continue for at least two months, five half-lives, after the last dose on study medication.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Prados MD, Schold SC Jr, Fine HA, Jaeckle K, Hochberg F, Mechtler L, Fetell MR, Phuphanich S, Feun L, Janus TJ, Ford K, Graney W. A randomized, double-blind, placebo-controlled, phase 2 study of RMP-7 in combination with carboplatin administered intravenously for the treatment of recurrent malignant glioma. Neuro Oncol. 2003 Apr;5(2):96-103. doi: 10.1093/neuonc/5.2.96. PMID 12672281
- [Background] Prados MD, Warnick RE, Mack EE, Chandler KL, Rabbitt J, Page M, Malec M. Intravenous carboplatin for recurrent gliomas. A dose-escalating phase II trial. Am J Clin Oncol. 1996 Dec;19(6):609-12. doi: 10.1097/00000421-199612000-00016. PMID 8931682
- [Result] A randomized phase II trial of Vandetanib (ZD6474) in combination with carboplatin versus carboplatin alone in adults with recurrent glioblastoma. Katherine McNeill, Fabio Iwamoto, Teri Kreisl, Joohee Sul, Joanna Shih, Howard Fine, New York University, New York, NY, USA, Columbia University, New York, NY, USA, National Institutes of Health, Bethesda, MD, USA, Food and Drug Administration, Silver Spring, MD, USA.
- [Result] A randomized phase II trial of Vandetanib in combination with carboplatin versus carboplatin alone followed by Vandetanib aline in adults with recurrent anaplastic astrocytoma. Prakash Ambady, Katherine Warren, Joanna Shih, Teri Kreisl, Howard Fine, National Institutes of Health, Bethesda, MD, USA.
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0222.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Vandetanib With Carboplatin: ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
  Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
Period: Overall Study
Arm/Group | Carboplatin | Vandetanib With Carboplatin
Started | 56 | 56
Crossover to Vandetanib | 42 | 0
Completed | 39 | 54
Not Completed | 17 | 2
Not completed — Withdrew consent | 1 | 0
Not completed — Refused further treatment | 8 | 2
Not completed — Toxicity | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin | Vandetanib With Carboplatin | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 105
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.29 (13.29) | 50.10 (12.43) | 50.13 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 37 | 41 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 55 | 56 | 111
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 53 | 52 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 112

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at 6 Months
Description: Percentage of participants who are alive and progression-free at 6 months.
Time Frame: 6 months
Population: The group data is displayed per the report provided to the Food and Drug Administration.
Measure: Number; unit: percentage of participants
Groups:
- Glioblastoma (Combination); Anaplastic Astrocytomas (Combination): ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
  Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
- Glioblastoma (Carboplatin Alone); Anaplastic Astrocytomas (Carboplatin Alone): Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
Arm/Group | Glioblastoma (Combination) | Glioblastoma (Carboplatin Alone) | Anaplastic Astrocytomas (Combination) | Anaplastic Astrocytomas (Carboplatin Alone)
Number analyzed (Participants) | 33 | 33 | 23 | 23
percentage of participants | 1.71 | 0.89 | 8.7 | 17.4

2. Secondary Outcome: Overall Survival
Description: Time between the first day of treatment and the day of death.
Time Frame: Time between the first day of treatment and the day of death, up to 1.5 years
Population: The group data is displayed per the report provided to the Food and Drug Administration.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Glioblastoma (Carboplation Alone); Anaplastic Astrocytoma (Carboplatin Alone): Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
- Anaplastic Astrocytoma (Combination): ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
  Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
Arm/Group | Glioblastoma (Combination) | Glioblastoma (Carboplation Alone) | Anaplastic Astrocytoma (Combination) | Anaplastic Astrocytoma (Carboplatin Alone)
Number analyzed (Participants) | 33 | 33 | 23 | 23
Months | 5.58 [4.60 to 8.65] | 5.22 [3.78 to 7.46] | 6.5 [5.42 to 11.7] | 9.27 [5.52 to 43.86]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 70 months and 19 days
Measure: Number; unit: participants
Groups:
- Carboplatin: Combo Group (both drugs together)
  ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
  Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
- Vandetanib With Carboplatin: Sequential Group (carboplatin followed by vandetanib)
  ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
  Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
- Cross Over to Vandetanib: ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
  Carboplatin: Carboplatin is a drug that interrupts division of cancer cells and has been shown to be a useful drug in treatment of tumors known as gliomas. It is a useful drug for treating brain tumors, but researchers are interested in gathering more information about how it works as a treatment for patients who have not responded to initial surgery, radiation, or chemotherapy.
Arm/Group | Carboplatin | Vandetanib With Carboplatin | Cross Over to Vandetanib
Number analyzed (Participants) | 56 | 56 | 42
participants | 55 | 56 | 40

ADVERSE EVENTS:
Groups:
- Crossover to Vandetanib: ZD6474 (Vandetanib): Vandetanib is an oral medication known to block angiogenesis and has shown significant antitumor activity in laboratory and animal studies. Vandetanib appears to be well tolerated by patients at specific daily doses.
Arm/Group | Carboplatin | Vandetanib With Carboplatin | Crossover to Vandetanib
Serious Adverse Events (participants affected / at risk) | 10/56 | 21/56 | 13/42
Other Adverse Events (participants affected / at risk) | 55/56 | 56/56 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin (N=56) | Vandetanib With Carboplatin (N=56) | Crossover to Vandetanib (N=42)
Death Not otherwise specified (NOS) (General disorders) | 1 (1) | 2 (2) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 1 (3) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 2 (3) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (UTI) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 4 (4) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (cellulitis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin (N=56) | Vandetanib With Carboplatin (N=56) | Crossover to Vandetanib (N=42)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 5 (11) | 1 (1)
Alanine aminotransferase increased (Investigations) | 19 (29) | 43 (74) | 24 (29)
Alkaline phosphatase increased (Investigations) | 4 (4) | 17 (20) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 30 (67) | 26 (74) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 28 (44) | 14 (17)
Blood bilirubin increased (Investigations) | 2 (2) | 8 (11) | 3 (3)
Cardiac disorders - Other, specify (Qtc prolonged) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (2) | 0 (0) | 3 (3)
Concentration impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 20 (40) | 12 (13)
Cushingoid (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 4 (4) | 3 (3) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 3 (5) | 22 (38) | 18 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (diplopia) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Stye) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 16 (29) | 19 (24) | 3 (3)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (cholelithiasis) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (sore throat) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 2 (3) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — aphasia and right upper extremity weakness
Nervous system disorders - Other, specify (visual field deficit) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 4 (5) | 2 (3) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 35 (45) | 24 (27)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — lung infection
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 7 (9) | 14 (33) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 3 (4) | 4 (4) | 5 (7)
Skin infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (6) | 1 (1)
Weight loss (Investigations) | 2 (2) | 6 (7) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 33 (108) | 29 (96) | 14 (17)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Acoustic nerve disorder Not otherwise specified (NOS) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (4) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 3 (5) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6) | 3 (4) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7) | 4 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (5) | 9 (11) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 6 (15) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 12 (23) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (7) | 15 (19) | 4 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 4 (8) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (9) | 17 (44) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (7) | 11 (14) | 5 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 19 (25) | 19 (34) | 11 (12)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (vaginal candidiasis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Had UTI with pseudomonas
Injury, poisoning and procedural complications - Other, specify (left shoulder fracture) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1) — Azotemia/Urea nitrogen (BUN)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 39 (122) | 44 (122) | 27 (44)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (11) | 9 (11) | 3 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — left side Hemineglect
Neutrophil count decreased (Investigations) | 18 (59) | 15 (48) | 5 (6)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (10) | 6 (6)
Platelet count decreased (Investigations) | 48 (119) | 51 (129) | 17 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (erythema) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 29 (46) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6) | 1 (1)
Headache (Nervous system disorders) | 8 (10) | 5 (6) | 4 (6)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 3 (3)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 23 (35) | 12 (14)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0)
Investigations - Other, specify (elevated LDH) (Investigations) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (2) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — elevated bilirubin
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — subdural hygroma
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 5 (8) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — nasal septum erosions
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Bug bites
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Morphea vs. psoriasiform plaque-left arm
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) — Sebaceous cyst
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Seborrheic dermatitis vs. inverse psoriasis-buttocks
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — skin laceration
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Inflammation around nail bed
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Navel area irritation
Skin and subcutaneous tissue disorders - Other, specify (paronychia) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — 2 reddened areas

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No